CLINICAL TRIAL: NCT04376710
Title: Surgical Telemedicine in the COVID-19 Pandemic Era
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 20-1177
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: COVID; Surgery
Keywords: Telemedicine; COVID; Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgeons
  Interventions: Other: Completion of pre-pandemic survey; Other: Completion of survey after peak of pandemic
- Patients
  Interventions: Other: Completion of post telemedicine encounter survey

INTERVENTIONS:
Other: Completion of pre-pandemic survey — Surgeons will take a pre-pandemic survey to determine surgeon perceptions to telemedicine and barriers to implementation.
  Groups: Surgeons
Other: Completion of survey after peak of pandemic — Surgeons will take another survey after the peak of pandemic to determine surgeon perceptions to telemedicine and barriers to implementation.
  Groups: Surgeons
Other: Completion of post telemedicine encounter survey — Patients will take a post telemedicine encounter survey to determine patient perceptions to telemedicine and barriers to implementation.
  Groups: Patients

SUMMARY:
The current COVID-19 pandemic has caused delays in initial or follow-up encounters between surgical patients and physicians. While this delay allows for resource allocation to those most severely affected by the pandemic, surgeons are faced with potential important delays in diagnosis and the expanding backlog of elective cases and initial evaluations.

This project will assess surgeon and patient telemedicine perspectives. Pre-pandemic views on telemedicine among a cohort of surgeons will be obtained and compared to views at 3 months from the peak of the pandemic. Patients will be surveyed following telemedicine appointments with an anonymous questionnaire to learn about patient receptiveness to telemedicine. Barriers to implementation will be addressed throughout the duration of the study.

ELIGIBILITY:
Inclusion Criteria

1. Surgical faculty at participating institutions will receive surveys regarding telemedicine early in the start of the study to assess baseline perceptions. These same group of surgeons will receive subsequent surveys 3 months after the peak of the pandemic to evaluate telemedicine perceptions following a rapid implementation and adoption of telemedicine.
2. Surgical patients evaluated from the start of the study through a 6-month period will be included in the study. They will have the option after each telemedicine encounter to complete an anonymous survey regarding perceptions to this technology.

Exclusion Criteria

1. No exclusions for surgical faculty are identified. Accrual of data from this group will be limited only by response rates to administered surveys.
2. Exclusions for surgical patients will include the inability to access the technology required for a telemedicine consultation (e.g.: absence of a camera enabled smartphone, absence of a required internet or cellular connection to perform a telemedicine encounter). The investigators will keep a list of reasons for the inability to perform a telemedicine encounter to identify the barriers to implementation among patients.

Ages: 31 Days to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Surgical faculty at participating institutions will be able to complete pre and post pandemic surveys regarding telemedicine and barriers to implementation.
  Surgical patients who complete a telemedicine encounter from the start of the study through a 6-month period will be included in the study. They will be able to complete an optional anonymous survey regarding perceptions to telemedicine and perceived barriers to implementation.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Evaluate surgeon perceptions to telemedicine and perceived barriers to implementation | 6 months
  Surgeons will take an anonymous survey early after the start of the study regarding perceptions to telemedicine and perceived barriers to implementation. Surgeons will be asked again after 3 months from the peak of the pandemic to take another survey to assess how the pandemic has changed perceptions to telemedicine and the observed barriers to implementation.
Evaluate patient perceptions to telemedicine and perceived barriers to implementation | 6 months
  Patients will take an optional anonymous survey at the end of each telemedicine encounter to assess patient perceptions to telemedicine and barriers to implementation.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
No plan for IPD.

REFERENCES:
- [Derived] Diaz-Miron J, Ogle S, Kaizer A, Acker SN, Rove KO, Inge TH. Surgeon, patient, and caregiver perspective of pediatric surgical telemedicine in the COVID-19 pandemic era. Pediatr Surg Int. 2022 Feb;38(2):241-248. doi: 10.1007/s00383-021-05016-8. Epub 2021 Sep 22. PMID 34550442